CLINICAL TRIAL: NCT06981299
Title: A Phase 1, First-In-Human, Randomized, Double-Blind, Placebo-Controlled Multi-Part Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of PROT-001, the Effect of Food and Age on the Pharmacokinetics of PROT-001, and the Effect of PROT-001 on the Pharmacokinetics of Digoxin and Rosuvastatin in Healthy Adult Participants.
Brief Title: A Phase 1 Study of PROT-001.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protego Biopharma Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Protego Biopharma, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO-1A-101
Record Dates: First submitted 2025-05-06; First posted 2025-05-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; Digoxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- SIngle ascending dose (Placebo Comparator): Part 1 is a randomized, double-blind, placebo-controlled study to evaluate single ascending doses of PROT-001 in healthy adult participants. Up to 7 sequential cohorts (including 6 planned and 1 optional dose level) of approximately 8 participants each (6 receiving PROT-001 and 2 receiving placebo), will be initiated. The planned dose levels of PROT-001 are tentative, with the first 2 dose levels planned at 15 mg and 75 mg. Subsequent cohorts will have dose levels increased by no more than 3-fold of the previous evaluated dose with the maximum dose not exceeding a single dose of 1800 mg during Part 1 of the study.
  Interventions: Drug: PROT-001
- Multiple ascending dose (Placebo Comparator): Part 2 is a randomized, double-blind, placebo-controlled study to evaluate multiple ascending doses of PROT-001 in healthy adult participants. Up to 3 sequential cohorts of approximately 8 participants each (6 receiving PROT-001 and 2 receiving placebo), will be enrolled. Tentative doses between 600 and 1800 mg administered twice daily (BID) for 14 days will be explored, with a maximum dose not exceeding 3600 mg/day. The exact multiple dosing frequency (i.e., BID or once daily [QD]) will be determined based on the estimated half-life, PD, and safety data following the single doses evaluated in Part 1. The maximum dose for the first MAD cohort will be the BID dosing of the highest SAD dose deemed to be safe and well tolerated by the SRC.
  Interventions: Drug: PROT-001
- Food-effect (Other): The Food-Effect arm is a randomized, open-label, 2-sequence, 2-period crossover, single-dose study to evaluate the effect of food on the PK of PROT-001 in 12 healthy adult participants. The proposed dose level will be a dose of PROT-001 that is deemed to be safe and well tolerated following single-dose administration, as determined following SRC review.
  Interventions: Drug: PROT-001
- Optional Age-effect (Other): The optional Age-Effect arm is an open-label, non-randomized, single-dose study to evaluate the effect of age on the PK of PROT-001 in healthy elderly participants (>65 to 75 years of age). The proposed dose level will be a dose of PROT-001 that is deemed to be safe and well tolerated following single-dose administration, as determined following SRC review.
  Interventions: Drug: PROT-001
- Drug-drug interaction (Other): The Drug-drug Interaction arm is a nonrandomized, open-label, 2-period, single sequence, DDI study to evaluate the potential interaction of PROT-001 on the PK of a 2-drug cocktail probe containing digoxin (a substrate of P-gp) and rosuvastatin (a substrate of BCRP, OATP1B1, and OATP1B3 transporters) in healthy adult participants. The proposed PROT-001 dose level will be a dose of PROT-001 that has been deemed to be safe and well tolerated from Part 2 (MAD) of the study.
  Interventions: Drug: PROT-001; Drug: Rosuvastatin 10mg; Drug: Digoxin 0.25 mg

INTERVENTIONS:
Drug: PROT-001 — Orally bioavailable small molecule kinetic stabilizer of lambda light chains (λLCs).
Drug: Rosuvastatin 10mg — A substrate of BCRP, OATP1B1, and OATP1B3 transporters
  Arms: Drug-drug interaction
Drug: Digoxin 0.25 mg — A substrate of P-gp
  Arms: Drug-drug interaction

SUMMARY:
A Phase 1, First-In-Human, Randomized, Double-Blind, Placebo-Controlled Multi-Part Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of PROT-001, the Effect of Food and Age on the Pharmacokinetics of PROT-001, and the Effect of PROT-001 on the Pharmacokinetics of Digoxin and Rosuvastatin in Healthy Adult Participants.

DETAILED DESCRIPTION:
This study will enrol approximately 122 participants, in four parts:

Part 1 is a single ascending (increasing) dose (SAD) study, where approximately 56 participants will receive a single dose of the study drug or placebo.

Part 2 is a multiple ascending (increasing) dose (MAD) study, where approximately 24 participants will receive multiple doses of the study drug or placebo for up to 14 days.

Part 3 is a food effect (FE) and age effect (AE) study, where approximately 12 participants in the food effect part of the study will receive 2 doses of the study drug: 1 dose after avoiding food for a set amount of time (fasted state), and 1 dose immediately after consuming a meal (fed state). Approximately 10 participants in the optional age effect part of the study will receive a single dose of the study drug after avoiding food for a set amount of time (fasted state).

Part 4 is a nonrandomized, open-label, 2-period, single sequence, DDI study to evaluate the potential interaction of PROT-001 on the PK of a 2-drug cocktail probe containing digoxin (a substrate of P-gp) and rosuvastatin (a substrate of BCRP, OATP1B1, and OATP1B3 transporters) in healthy adult participants. The proposed PROT-001 dose level will be a dose of PROT-001 that has been deemed to be safe and well tolerated from Part 2 (MAD) of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of providing written, signed, and dated participant informed consent prior to any study-related procedures, as described in Section 10.1.4.
2. For all study parts except Part 3 (Age-Effect study), participants must be between 18 and 65 years of age (inclusive) at the time of Screening (signing the ICF). For Part 3 (Age-Effect study) only, participants must be >65 to 75 years of age at the time of Screening.
3. Has a body mass index (BMI) of 18 to 32 kg/m2 (inclusive) and a body weight of ≥50 kg.
4. Is judged by the Investigator to be generally healthy, as determined by a medical history without major pathology, and no clinically significant findings based on physical examination, 12-lead electrocardiogram (ECG), vital signs, and clinical laboratory results obtained at Screening and on days of admission to the study site (Day -1 and Day 14, as appropriate).
5. For all study parts except Part 3 (Age-Effect study), estimated glomerular filtration rate (eGFR) must be >90 mL/min/1.73 m2 at Screening; for Part 3 (Age-Effect study), eGFR must be ≥60 mL/min/1.73 m2 (using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine Equation [2021]).
6. Has a resting pulse (after at least 5 minutes of rest) within the following ranges:

   1. Parts 1 to 3: 40 to 100 beats per minute
   2. Part 4: 50 to 100 beats per minute

   Systolic and diastolic blood pressure (BP) must be 90-140/40-90 mmHg for all parts of the study.
7. Participants assigned female at birth are eligible to participate if they are not pregnant, not breastfeeding, and at least ONE of the following conditions applies:

   * Are a participant of nonchildbearing potential:
   * Surgically sterile (documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy), or
   * Are postmenopausal (amenorrhea for ≥12 months without an alternative medical cause AND a follicle-stimulating hormone [FSH] level >40 IU/L), or
   * Is a woman of childbearing potential (WOCBP) and agree to have their partner use a condom, and, if their partner is not vasectomized (with documented azoospermia), to use a highly effective method of contraception consistently and correctly starting from 1 month prior to Screening until at least 45 days after the last dose of IP.
8. Participants assigned male at birth who are sexually active with a female partner of childbearing potential are eligible to participate if they agree to use a condom, and have either been vasectomized (with documented azoospermia) or agree to have their partner use a highly effective method of contraception from Day 1 until at least 105 days after the last dose of IP.
9. Participants must refrain from donating eggs (ova, oocytes) from Day 1 until at least 45 days or sperm from Day 1 until at least 105 days after receiving the last dose of the IP.
10. Participants, who, in the opinion of the Investigator, can and will comply with the requirements and restrictions, including lifestyle restrictions listed in the Protocol.
11. Able to swallow an oral solid-dosage form of medication.
12. For Part 3 (Food-Effect study) only, able to consume a standardized high-fat meal.

Exclusion Criteria:

1. History or current evidence of a clinically significant or uncontrolled underlying condition, including but not limited to cardiovascular, hepatic, renal, hematological, infectious, autoimmune, neurological, psychiatric, endocrine, gastrointestinal, reproductive, pulmonary, or ocular. Clinically significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the participant at risk through participation or which could affect the endpoint analysis if the disease/condition worsened during the study.

   EXCEPTION: Fully resolved childhood asthma is not exclusionary. Note: In Part 3 Age-Effect study, participants with well-controlled non-serious chronic medical conditions managed by permitted medications (e.g. chronic asthma, hypertension, dyslipidemias) may be enrolled according to PI judgment, in consultation with the Medical Monitor if required.
2. History of or current invasive malignancy including hematological malignancies. Participants with a history of basal cell or squamous cell carcinoma or other carcinomas in situ that has been treated with no evidence of recurrence within 1 year prior to Screening will be allowed for inclusion, as judged by the Investigator.
3. History or presence of any disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
4. Any current active infections, including localized infections, or any recent history of active infections, cough, or fever within 1 week prior to IP administration (including severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2]), or any history of recurrent or chronic infections.
5. Known history of significant multiple and/or severe allergies (e.g., food, drug, or latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e., systemic allergic reaction) to prescription or nonprescription drugs or food. EXCEPTION: Untreated, asymptomatic, seasonal allergies are not exclusionary.
6. Family history of sudden death or of congenital prolongation of the QT interval corrected for heart rate (QTc) or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval.
7. Known or suspected hypersensitivity to any component of the finished dosage form of PROT-001.
8. Tested positive for hepatitis B surface antigen, anti-hepatitis C virus antibodies, or anti-human immunodeficiency virus 1 and 2 antibodies at Screening.
9. In the 12-lead ECG assessment at Screening or on days of admission to the study site (Day -1 and Day 14, as appropriate), QTcF >450 msec. NOTE: One repeat screen is allowed at the discretion of the Investigator.
10. Has absolute neutrophil count (ANC) <2 × 109/L or aspartate transaminase (AST) and alanine transaminase (ALT) >1.5 × ULN, or INR >1.2 at Screening or on days of admission to the study site (Day -1 and Day 14, as appropriate).
11. Has positive urine drug (excluding positive for cotinine) or alcohol breath test results at Screening or on days of admission to the study site (Day -1 and Day 14, as appropriate).
12. Use of more than 10 tobacco nicotine-containing products (e.g., 10 cigarettes) per week within 3 months prior to the first IP administration and should agree to follow the restrictions related to tobacco/nicotine-containing consumption during the study, as outlined in the Protocol.
13. Any history of alcohol abuse, with an average intake exceeding 21 drinks per week for men, 14 drinks per week for women, or >4 drinks in 1 sitting several times a week (1 drink is equivalent to 12 g alcohol [i.e., 150 mL of wine, 360 mL of beer, or 45 mL of 80-proof distilled spirits]) or drug addiction (including soft drugs like cannabis products).
14. Use of any prescription or non-prescription medications, including over-the-counter (OTC) medications, vitamins, multivitamins, recreational drugs, dietary supplements, and herbal remedies such as St. John's Wort extract, or drugs considered likely to interfere with the safe conduct of the study within 7 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of the IP, or their planned use during the study period. EXCEPTIONS: After randomization, ibuprofen (≤1.2 g in 24 hours) and/or paracetamol (≤4 g in 24 hours but ≤1 g in 4 hours) may be administered at the discretion of the Investigator or delegate. Thyroid hormone replacement medication may be permitted if the participant has been on same stable dose for the last 3 months prior to the first dose of IP. Hormone replacement therapy and hormonal contraceptives will also be allowed.
15. Received an investigational drug within 30 days or 5 half-lives (whichever is greater) prior to the first dose of IP.
16. Has received any live vaccines (bacterial or viral) within 30 days prior to the first dose of IP or intend to receive a live vaccine during the study period.

    EXCEPTIONS: Vaccines allowed by the protocol include inactivated flu and COVID-19 vaccines in all participants. The recommended time intervals for administration of these vaccines are at least 7 days before the first dose of IP or 7 days after the last dose of IP.
17. Plans to donate or has donated ≥350 mL of blood (including blood products) within 28 days prior to the first dose of IP.
18. Plans to donate or has donated plasma within 7 days prior to the first dose of IP.
19. Female participant who is pregnant, breastfeeding, or plans to become pregnant or donate ova for in vitro fertilization during the study period and for 45 days following the last dose of IP or male participant who plans to donate sperm for in vitro fertilization during the study period and for 105 days following the last dose of IP.
20. The participant is considered to be vulnerable (e.g., cognitively impaired, or a person kept in detention).
21. The participant is an employee of the study site or has a family member or household member involved with the conduct of this study.
22. Any reason that in the opinion of the Investigator would lead to the inability of the participant to comply with the protocol.
23. Part 4 only: Known or suspected hypersensitivity to digoxin and/or rosuvastatin, their excipients, or any contraindication to their use.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Safety Outcome Measures (Adverse Events) | From enrollment through 6 weeks for SAD participants, 7 weeks for MAD participants, and 7 weeks for Food Effect and Age Effect participants.
  Occurrence of adverse events (AEs) of any type and severity.
Safety outcome measures (Vital signs: Systolic Blood Pressure) | From enrollment through 6 weeks for SAD participants, 7 weeks for MAD participants, and 7 weeks for Food Effect and Age Effect participants.
  SBP will be measured in mmHg
Safety outcome measures (Vital signs: Heart Rate) | From enrollment through 6 weeks for SAD participants, 7 weeks for MAD participants, and 7 weeks for Food Effect and Age Effect participants.
  Heart rate will be measured in bpm
Safety outcome measures (Vital signs: Respiratory Rate) | From enrollment through 6 weeks for SAD participants, 7 weeks for MAD participants, and 7 weeks for Food Effect and Age Effect participants.
  Heart rate will be measured in rpm
Safety outcome measures (Vital signs: Temperature) | From enrollment through 6 weeks for SAD participants, 7 weeks for MAD participants, and 7 weeks for Food Effect and Age Effect participants.
  Body temperature will be measured in Celsius (0C)
Safety outcome measures (ECG QTCF Interval) | From enrollment through 6 weeks for SAD participants, 7 weeks for MAD participants, and 7 weeks for Food Effect and Age Effect participants.
  The QTcF interval will be calculated using the formula QTcF = QT/√R-R interval in seconds.
Safety outcome measures (Clinical Laboratory Parameters) | From enrollment through 6 weeks for SAD participants, 7 weeks for MAD participants, and 7 weeks for Food Effect and Age Effect participants.
  For parameters outside of the reference range an assessment of the significance (clinically significant / non-clinically significant) will be provided and all data outside the reference range of the clinical laboratory will be listed for all study participants.
Safety Outcome Measures (Physical Exam) | From enrollment through 6 weeks for SAD participants, 7 weeks for MAD participants, and 7 weeks for Food Effect and Age Effect participants.
  Occurrence of abnormal clinically significant finding on physical examination as assessed by the Investigator.
Part 4 - Pharmacokinetics Outcome Measures (Cmax) | At steady state (Day 12), compared to baseline values obtained prior to PROT-001 administration (Day 1).
  The maximum concentration achieved by PROT-001, digoxin and rosuvastatin following administration of PROT-001
Part 4 - Pharmacokinetics Outcome Measures (AUC(0-inf)) | At steady state (Day 12), compared to baseline values obtained prior to PROT-001 administration (Day 1).
  Area under the concentration achieved by PROT-001, digoxin and rosuvastatin following administration of PROT-001. Reflects the actual body exposure to drug after administration of a dose of the drug and is expressed in mg*h/L.

SECONDARY OUTCOMES:
Pharmacokinetics Outcome Measures (Cmax) | Day 1 for the SAD, Food Effect and Age Effect parts and Days 1 and 14 for the multiple dosing parts.
  The maximum concentration achieved by PROT-001 in a specified compartment area of the body after the drug has been administered and before the administration of a second dose.
Pharmacokinetics Outcome Measures (Tmax) | Day 1 for the SAD, Food Effect and Age Effect parts and Days 1 and 14 for the multiple dosing parts. Days 1 and 12 for Part 4 DDI.
  Time at which maximum concentration of PROT-001 is reached
Pharmacokinetics Outcome Measures (half-life (t1/2)) | Day 1 for the SAD, Food Effect and Age Effect parts and Days 1 and 14 for the multiple dosing parts. Days 1 and 12 for Part 4 DDI.
  The estimate of the time it takes for the concentration or amount in the body of that drug to be reduced by exactly one-half (50%).
Pharmacokinetics Outcome Measures (AUC0-t and AUC0-inf) | Day 1 for the SAD, Food Effect and Age Effect parts and Days 1 and 14 for the multiple dosing parts. Days 1 and 12 for Part 4 DDI.
  Area under the concentration curve (AUC0-t and AUC0-inf) reflects the actual body exposure to drug after administration of a dose of the drug and is expressed in mg*h/L.
Pharmacokinetics Outcome Measures (Total Plasma Clearance (CL)) | Day 1 for the SAD, Food Effect and Age Effect parts and Days 1 and 14 for the multiple dosing parts. Days 1 and 12 for Part 4 DDI.
  The volume of drug cleared from blood or plasma in unit time.
Pharmacokinetics Outcome Measures (Volume of Distribution (Vd)) | Day 1 for the SAD, Food Effect and Age Effect parts and Days 1 and 14 for the multiple dosing parts. Days 1 and 12 for Part 4 DDI.
  PROT-001's propensity to either remain in the plasma or redistribute to other tissue compartments.
Pharmacodynamics Outcome Measures (Light Chain (LC) Stabilization) | From enrollment through Day 3 for SAD participants, through day 16 for MAD participants, through Day 3 for Age Effect participants.
  Confirmation of target engagement, in terms of LC stabilization in plasma, using the AmyLite™ assay.
Part 4 - Safety outcome measures (Adverse Events) | From enrollment through Day 23.
  Occurrence of adverse events (AEs) of any type and severity.
Part 4 - Safety outcome measures - Number of participants with abnormal Clinical Laboratory Parameters) | From enrollment through Day 23.
  For parameters outside of the reference range an assessment of the significance (clinically significant / non-clinically significant) will be provided and all data outside the reference range of the clinical laboratory will be listed for all study participants.
Part 4 - Safety outcome measures (Vital signs - Respiratory Rate) | From enrollment through Day 23.
  Heart rate will be measured in rpm
Part 4 - Safety outcome measures (Vital signs - Respiratory Rate) | From enrollment through Day 23.
  Respiratory rate will be measured in rpm
Part 4 - Safety outcome measures (Vital signs - Temperature) | From enrollment through Day 23.
  Temperature will be measured in Celsius (0C)
Part 4 - Safety outcome measures (ECG QTCF Interval) | From enrollment through Day 23.
  The QTcF interval will be calculated using the formula QTcF = QT/√R-R interval in seconds.
Part 4 - Safety outcome measures (Physical Exam) | From enrollment through Day 23.
  Occurrence of abnormal clinically significant finding on physical examination as assessed by the Investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia